CLINICAL TRIAL: NCT05359614
Title: A Single-centered Randomized Single-blinded Clinical Trial to Evaluate Efficacy and Safety of Sequential Treatment of CoolSculpting Elite With CoolTone vs. CoolSculpting Elite Alone in Treating the Banana Roll Region
Brief Title: Coolsculpting With Cooltone Verses Coolsculpting Alone for the Banana Roll Area
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Coolsculpt-Cooltone-2022
Record Dates: First submitted 2022-03-18; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Improved Appearance of the Banana Roll Region

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- GROUP A=CoolSculpting Elite and CoolTone (Experimental): Group A: Study subjects will have a total of 1 or 2 bilateral CoolSculpting Elite sessions to the banana roll area 6 weeks prior to four EMMS treatment sessions during the study.
  Interventions: Device: CoolSculpting Elite combined with CoolTone Treatments
- GROUP B CoolSculpting Elite alone (Active Comparator): Group B: Study subjects will have a total of 1 or 2 bilateral CoolSculpting Elite sessions to the banana roll area.
  Interventions: Device: CoolSculpting Elite

INTERVENTIONS:
Device: CoolSculpting Elite combined with CoolTone Treatments — Coolsculpting treatment combined with Cooltone treatments for the banana roll region of the buttocks.
  Arms: GROUP A=CoolSculpting Elite and CoolTone
Device: CoolSculpting Elite — Coolsculpting treatment alone for the banana roll region of the buttocks
  Arms: GROUP B CoolSculpting Elite alone

SUMMARY:
to evaluate the benefit and efficacy of CoolSculpting Elite study treatments versus CoolSculpting Elite study treatments followed by a series CoolTone for underneath the buttocks (also known as the banana roll).

DETAILED DESCRIPTION:
Investigate safety and efficacy of CoolSculpting Elite treatments for underneath the buttocks (also known as the banana roll) versus sequential treatments of CoolSculpting Elite and CoolTone for the banana roll region.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  1. Female ≥ 22 years and ≤65 years of age.
  2. Subject has not had weight change exceeding 5% of body weight in the preceding month.
  3. Subject agrees to maintain body weight within 5% during the study by not making any changes in diet or exercise routine.
  4. Subject has a BMI ≤ 30 as determined at screening.
  5. Subject agrees to have photographs taken of the treatment area(s) during the scheduled time periods.
  6. Subject agrees to refrain from any new or change in gluteal muscle training exercises of the treatment area during the course of the study.
  7. Subject agrees to avoid sun tanning or spray tanning during the course of the study. Subject has read and signed the study written informed consent form

Exclusion Criteria:

* Exclusion Criteria

  1. Male Subjects
  2. Subject has had a recent surgical procedure(s) in the area of intended treatment and muscle contractions may disrupt the healing process.
  3. A subject with any uncontrolled systemic disease. A potential subject in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study.
  4. A subject with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
  5. Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) non-invasive fat reduction or skin tightening procedures , or cellulite treatment in the area of intended treatment
  6. Subjects who tanned or spray tanned in the treatment area within the past 4 weeks
  7. A subject with history of or the presence of any skin condition/disease in the treatment area that might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, eczema, psoriasis, seborrheic dermatitis) at the discretion of the investigator.
  8. Subject needs to administer or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month
  9. Subject hashad an intrauterine contraceptive device inserted or removed within the past month.
  10. A subject with an active bacterial, fungal, or viral infection in the treatment area.
  11. Subject has a bleeding disorder
  12. Subject has a blood disorder such as cryoglobulinemia, cold agglutinin disease and paroxysmal cold hemoglobinuria.
  13. Known sensitivity to cold such as cold urticaria, Raynaud's disease, pernio or Chilblains. Or patients with any impaired sensation in treated area
  14. A subject with scarring or tattoos in the treatment area that might interfere with the diagnosis or study evaluations at the discretion of the investigator.
  15. Subject is taking or has taken diet pills or supplements within the past month.
  16. Subject has a metal implant or active implanted device such as a cardiac pacemaker, cochlear implant, intrathecal pump, hearing aids, defibrillator, or drug delivery system.
  17. Subject has pulmonary insufficiency.
  18. Subject has a cardiac disorder.
  19. Subject has a malignant tumor.
  20. Subject has been diagnosed with a seizure disorder such as epilepsy.
  21. Subject currently has a fever.
  22. Subject is diagnosed with Grave's disease.
  23. Subject is pregnant or intending to become pregnant during the study period (in the next 9 months).
  24. Subject is lactating or has been lactating in the past 6 months.
  25. Subject is unable or unwilling to comply with the study requirements.
  26. Subject is currently enrolled in a clinical study of any other investigational drug or device.
  27. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.
  28. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject

Ages: 22 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
appearance of the banana roll region based on Investigator Global Aesthetic Improvement Scales | baseline to 6-weeks
  Investigator Global Aesthetic Improvement Scale Scores will be assigned where -3 = Very Much Worse, -2 = Much Worse -, -1 = Worse, 0 = No Chance, 1 = Improved, 2 = Much Improved, 3 = Very Much Improved
appearance of the banana roll region based on Investigator Global Aesthetic Improvement Scales | baseline to 7-weeks
  Investigator Global Aesthetic Improvement Scale Scores will be assigned where -3 = Very Much Worse, -2 = Much Worse -, -1 = Worse, 0 = No Chance, 1 = Improved, 2 = Much Improved, 3 = Very Much Improved
appearance of the banana roll region based on Investigator Global Aesthetic Improvement Scales | baseline to 12-weeks
  Investigator Global Aesthetic Improvement Scale Scores will be assigned where -3 = Very Much Worse, -2 = Much Worse -, -1 = Worse, 0 = No Chance, 1 = Improved, 2 = Much Improved, 3 = Very Much Improved
appearance of the banana roll region based on Investigator Global Aesthetic Improvement Scales | baseline to 13-weeks
  Investigator Global Aesthetic Improvement Scale Scores will be assigned where -3 = Very Much Worse, -2 = Much Worse -, -1 = Worse, 0 = No Chance, 1 = Improved, 2 = Much Improved, 3 = Very Much Improved
appearance of the banana roll region based on Investigator Global Aesthetic Improvement Scales | baseline to 18-weeks
  Investigator Global Aesthetic Improvement Scale Scores will be assigned where -3 = Very Much Worse, -2 = Much Worse -, -1 = Worse, 0 = No Chance, 1 = Improved, 2 = Much Improved, 3 = Very Much Improved
Improvement in Appearance of the Banana Roll Region Based on Clinical Photographs | 18 Weeks
  Investigator Global Aesthetic Improvement Scale Scores where -3 = Very Much Worse, -2 = Much Worse -, -1 = Worse, 0 = No Chance, 1 = Improved, 2 = Much Improved, 3 = Very Much Improved will be assigned by a blinded assessor based on photographs

SECONDARY OUTCOMES:
Patient Treatment Satisfaction Survey | baseline to 1-Week
  Subject rating of treatment satisfaction where - 3 = Completely Dissatisfied, -2 = Moderately Dissatisfied, -1 = Mildly Dissatisfied, 0 = Neither Satisfied nor Dissatisfied, 1 = Mildly Satisfied, 2 = Moderately Satisfied, 3 =Completely Satisfied
Patient Treatment Satisfaction Survey | baseline to 6-weeks
  Subject rating of treatment satisfaction where - 3 = Completely Dissatisfied, -2 = Moderately Dissatisfied, -1 = Mildly Dissatisfied, 0 = Neither Satisfied nor Dissatisfied, 1 = Mildly Satisfied, 2 = Moderately Satisfied, 3 =Completely Satisfied
Patient Treatment Satisfaction Survey | baseline to 7-weeks
  Subject rating of treatment satisfaction where - 3 = Completely Dissatisfied, -2 = Moderately Dissatisfied, -1 = Mildly Dissatisfied, 0 = Neither Satisfied nor Dissatisfied, 1 = Mildly Satisfied, 2 = Moderately Satisfied, 3 =Completely Satisfied
Patient Treatment Satisfaction Survey | baseline to 12-weeks
  Subject rating of treatment satisfaction where - 3 = Completely Dissatisfied, -2 = Moderately Dissatisfied, -1 = Mildly Dissatisfied, 0 = Neither Satisfied nor Dissatisfied, 1 = Mildly Satisfied, 2 = Moderately Satisfied, 3 =Completely Satisfied
Patient Treatment Satisfaction Survey | baseline to 13-weeks
  Subject rating of treatment satisfaction where - 3 = Completely Dissatisfied, -2 = Moderately Dissatisfied, -1 = Mildly Dissatisfied, 0 = Neither Satisfied nor Dissatisfied, 1 = Mildly Satisfied, 2 = Moderately Satisfied, 3 =Completely Satisfied
Patient Treatment Satisfaction Survey | baseline to 18-weeks
  Subject rating of treatment satisfaction where - 3 = Completely Dissatisfied, -2 = Moderately Dissatisfied, -1 = Mildly Dissatisfied, 0 = Neither Satisfied nor Dissatisfied, 1 = Mildly Satisfied, 2 = Moderately Satisfied, 3 =Completely Satisfied
Subject Global Aesthetic Improvement Scale | baseline to 6-weeks
  Subject rating of treatment results where where -3 = Very Much Worse, -2 = Much Worse -, -1 = Worse, 0 = No Chance, 1 = Improved, 2 = Much Improved, 3 = Very Much Improved
Subject Global Aesthetic Improvement Scale | baseline to 7-weeks
  Subject rating of treatment results where where -3 = Very Much Worse, -2 = Much Worse -, -1 = Worse, 0 = No Chance, 1 = Improved, 2 = Much Improved, 3 = Very Much Improved
Subject Global Aesthetic Improvement Scale | baseline to 12-weeks
  Subject rating of treatment results where where -3 = Very Much Worse, -2 = Much Worse -, -1 = Worse, 0 = No Chance, 1 = Improved, 2 = Much Improved, 3 = Very Much Improved
Subject Global Aesthetic Improvement Scale | baseline to 13-weeks
  Subject rating of treatment results where where -3 = Very Much Worse, -2 = Much Worse -, -1 = Worse, 0 = No Chance, 1 = Improved, 2 = Much Improved, 3 = Very Much Improved
Subject Global Aesthetic Improvement Scale | baseline to 18-weeks
  Subject rating of treatment results where where -3 = Very Much Worse, -2 = Much Worse -, -1 = Worse, 0 = No Chance, 1 = Improved, 2 = Much Improved, 3 = Very Much Improved

CONTACTS AND LOCATIONS:
Locations (1):
- West Dermatology Research Center/Cosmetic Laser Dermatology, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided